CLINICAL TRIAL: NCT03757663
Title: UV Dosimetry Feedback in Non-Melanoma Skin Cancer Patients
Brief Title: UV Dosimetry Feedback in NMSC Patients
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Study closed
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 17-2134.cc
Record Dates: First submitted 2018-11-26; First posted 2018-11-29 (Actual); Last update posted 2019-09-06 (Actual); Status verified 2019-09

CONDITIONS: Non-Melanoma Skin Cancer
Keywords: UV Dosimetry; UV Exposure; Behavioral; Social Cognitive Theory; Self-Regulation; Self-Efficacy
MeSH Terms: conditions — Behavior; Self-Control

STUDY DESIGN:
Intervention Model Description: Each participant will self-report skin protective behaviors and attitudes before wearing a UV dosimeter for 3 weeks. After the wear period, the study team provides feedback based on UV exposure. The participant will then wear the device again for 3 weeks.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- UV Dosimeter (Experimental): UV Dosimeter will measure participants' UV exposure for two separate 3-week periods.
  Interventions: Behavioral: UV Counseling

INTERVENTIONS:
Behavioral: UV Counseling — Participants will self-report their knowledge and attitudes related to UV exposure. They will then wear a dosimeter for 3 weeks. After, the study team will counsel the participants on their UV levels and exposure, creating a personal plan and advice for avoiding sun exposure before letting the participants wear the dosimeter for an additional 3 weeks.

SUMMARY:
This study aims to characterize UV exposures among NMSC patients (those with a history of skin cancer) and to pilot an innovative behavioral intervention to decrease modifiable UV exposures. It will use UV dosimeters to objectively measure UV exposure and provide time and activity specific UV data on an individual level. These data will be used to develop a targeted and personalized behavioral feedback plan with counseling aimed at effective sun exposure behavior change

DETAILED DESCRIPTION:
The study will focus on helping to prevent NMSC and its associated morbidity through learning when patients are unintentionally exposed to extreme UV radiation. It will then help to create manageable and realistic behavioral interventions to reduce exposure, while also educating patients of the dangers of abundant sun exposure.

ELIGIBILITY:
Inclusion Criteria:

* Patients between ages 18 and 50.
* Must be diagnosed with non-melanoma skin cancer.

Exclusion Criteria:

* Patients, who at the discretion of the clinician, are too ill or sick.
* Non-English speaking patients.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2018-03-12 (Actual); Primary Completion 2019-08-30 (Actual); Study Completion 2019-08-30 (Actual)

PRIMARY OUTCOMES:
Identify Discrepancies of Self-Reported Sun Exposure and Actual Sun Exposure | Start of study to end of study, up to 3 months
  Measured using individual dosimeters and comparing it to what participants state they believe their level of sun exposure is
Identify Discrepancies of Self-Reported Sun Exposure and Actual Sun Exposure | Start of study to end of study, up to 3 months
  Compare specific sun exposure behaviors responsible for the level of exposure versus what could be done to lessen it

SECONDARY OUTCOMES:
Behavioral Intervention and immediate follow-up | Start of study to end of study, up to 3 months
  Participants will receive a personalized feedback plan and the success of the plan will be measured through individual dosimetry. We will track real time change in sun exposure based on repeat UV dosimetry.
Long Term Follow Up - longitudinal change in sun exposure based on dosimetry | Start of study to end of study, up to 3 months
  Track the longitudinal change in sun exposure comparing baseline UV dosimetry measurements to 3 month follow up dosimetry measurements to determine if the changes observed in outcome 3 are maintained.

CONTACTS AND LOCATIONS:
Overall Officials: Myles Cockburn, PhD, Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado, Aurora, Colorado, United States